CLINICAL TRIAL: NCT04767464
Title: Feasibility of Providing a Purpose Renewal Intervention for Cancer Survivors Via Virtual Groups
Acronym: CC-V
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mary Radomski (Other)
Responsible Party: Sponsor-Investigator, Mary Radomski, Senior Scientific Advisor, Allina Health System
Organization: Allina Health System (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CKRC2021-CCV
Record Dates: First submitted 2021-02-11; First posted 2021-02-23 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer; Breast Neoplasm
Keywords: Purpose
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Compass Course (Other): Virtual Compass Course
  Interventions: Other: Compass Course

INTERVENTIONS:
Other: Compass Course — The Compass Course is an 8-session group course designed to address purpose in life of those with Breast Cancer. Enrollment in this arm will involve participation in the Compass Course virtually.

SUMMARY:
The Compass Course (CC) is a group intervention designed for individuals with Breast Cancer. Over the course of 8 face-to-face group sessions, the CC is designed to help participants reclaim a sense of self-grounded purpose in daily life, defined as intentional use of time and energy in ways that align with one's values, strengths, and sources of personal meaning (e.g., inner compass) in the moments that compose a day. Because of COVID-19, in-person groups are discouraged and so we need to identify new ways to provide group-based interventions that are feasible and efficacious.

ELIGIBILITY:
Inclusion Criteria:

1. Able to attend intervention sessions for 9 weeks on Monday or Tuesday afternoons (4:30 - 6:30 pm) starting Monday, April 5, 2021
2. 25 years of age or older
3. Completed chemotherapy and/or radiation treatment for Stage 0, 1, 2, or 3 breast cancer at least 2 months prior to participating in the Compass Course intervention
4. English speaking
5. Graduated from high school
6. Able to see, hear, speak (with or without assistive devices)
7. Able to provide own transportation to sessions
8. Willing and able to commit to attend all 8 intervention sessions
9. Access to computer or tablet and adequate internet connection to participate in video conference

Exclusion Criteria:

1. Stage 4 breast cancer or any other cancer
2. Actively receiving chemotherapy or radiation treatments for cancer. (However, patients may be on Herceptin and/or endocrine treatment and participate in the study.)
3. History of neurologic disorder (such as stroke or brain injury) with residual impairments that likely interfere with learning
4. Any medical condition (physical or mental health) that interferes with the performance of everyday activities and roles.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
Change in Scales of Psychological Wellbeing | Through Study Completion (about 4 Months)
  A widely-used self-report questionnaire that was designed to measure 6 theoretically motivated dimensions of psychological well-being (autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, self-acceptance).
Change in Meaning in Life Questionnaire | Through Study Completion (about 4 Months)
  A 10-item questionnaire designed to measure 2 dimensions of meaning in life: Presence of Meaning (how much respondents feel their lives have meaning) and Search for Meaning (how much respondents strive to find meaning and understanding in their lives).
Change in Engagement in Meaningful Activities survey | Through Study Completion (about 4 Months)
  A 12-item self-report questionnaire designed to measure the extent to which a person experiences meaningfulness in his/her daily life activities.
Change in Purpose Status Question | Through Study Completion (about 4 Months)
  A single forced-choice self-report screener question that we developed in order to characterize existential distress related to purpose in life.

SECONDARY OUTCOMES:
Change in Beck Depression Inventory -- II | Through Study Completion (about 4 Months)
  A 21-question, widely-used self-report rating inventory that measures characteristic attitudes and symptoms of depression.
Change in State-Trait Anxiety Inventory | Through Study Completion (about 4 Months)
  A self-report questionnaire composed of 20 state and 20 trait statements related to anxiety. We will use the 20-item State inventory (1-4 scale).

CONTACTS AND LOCATIONS:
Overall Officials: Mary V Radomski, OTR/L, PhD, Principal Investigator — Senior Scientific Advisor
Locations (1):
- Abbott Northwestern Hospital, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No